CLINICAL TRIAL: NCT02118662
Title: Energy Expenditure During Seated, Seated Cycling, and Treadmill Walking Work Conditions (EE-Work)
Acronym: EE-Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Neil Johannsen, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PBRC 2013-033
Record Dates: First submitted 2014-03-26; First posted 2014-04-21 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Energy Expenditure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Male Cohort (Experimental): Eight Male participants per cohort will complete the following:
  Energy Expenditure during seated in an office chair during normal rest. Energy Expenditure during seated and typing. Energy Expenditure during Treadmill walking work condition. Energy Expenditure during cycling work condition
  Interventions: Other: Energy Expenditure during seated in an office chair; Other: Energy Expenditure during seated and typing; Other: Energy Expenditure during Treadmill walking work condition; Other: Energy Expenditure during cycling work condition
- Female Cohort (Experimental): Eight femalel participants per cohort will complete the following:
  Energy Expenditure during seated in an office chair during normal rest. Energy Expenditure during seated and typing. Energy Expenditure during Treadmill walking work condition. Energy Expenditure during cycling work condition
  Interventions: Other: Energy Expenditure during seated in an office chair; Other: Energy Expenditure during seated and typing; Other: Energy Expenditure during Treadmill walking work condition; Other: Energy Expenditure during cycling work condition

INTERVENTIONS:
Other: Energy Expenditure during seated in an office chair — You will first rest motionless in a chair for 20 minutes. You will complete the working conditions for 15 minutes each at your own self-selected level of effort. A rest period of 5 minutes will be given between each condition. During the working conditions, you will be asked to retype a displayed standard set of text.
Other: Energy Expenditure during seated and typing — You will complete this working conditions for 15 minutes. A rest period of 5 minutes will be given between each condition. During the working conditions, you will be asked to retype a displayed standard set of text.
Other: Energy Expenditure during Treadmill walking work condition — You will complete the working conditions for 15 minutes each at your own self-selected level of effort. A rest period of 5 minutes will be given between each condition. During the working conditions, you will be asked to retype a displayed standard set of text.
Other: Energy Expenditure during cycling work condition — You will complete the working conditions for 15 minutes each at your own self-selected level of effort. A rest period of 5 minutes will be given between each condition. During the working conditions, you will be asked to retype a displayed standard set of text.

SUMMARY:
The study is designed to measure the energy expenditure associated with a common office task (i.e., typing) while 1.) seated in an office chair, 2.) pedaling using a prototype pedal desk, and 3.) walking on a treadmill.

DETAILED DESCRIPTION:
The anthropometrics will be measured first. The height and body weight will be collected by clinic staff in the clinic.

The metabolic testing of all conditions will take place in a real office setting. The participant will be fitted with a heart rate monitor fastened around their chest using an elastic strap. They will also be fitted with a portable metabolic system (COSMED). This unit fits around their waist and back, much like a backpack. The unit is attached to a face mask that fits over their mouth and nose and is secured by elastic straps which wrap around their head.

The participants will first rest motionless in a chair for 20 minutes. Following this, they will complete three different simulated working conditions by typing at a computer while 1) seated in an office chair, 2) seated pedaling while using a prototype pedal desk, and 3) walking on a treadmill. The order of testing for the seated pedaling and treadmill walking working conditions will be counterbalanced with participants randomly assigned to the two possible order permutations. They will complete the 3 working conditions for 15 minutes each at their own self-selected level of effort. A rest period of 5 minutes will be given between each condition. During the working conditions, they will be asked to retype a displayed standard set of text.

ELIGIBILITY:
Inclusion Criteria:

* You are a full-time employee at the Pennington Biomedical Research Center
* You are between 21 and 65 years of age
* You previously participated in the Pennington Biomedical Research Center's Worker's Acceptability of a Prototype Integrated and Interactive Pedal Desk study (WAPD study)
* You are familiar with using word processing software and comfortable using a standard computer keyboard
* You primarily sit while at work

Exclusion Criteria:

* You weigh more than 250 pounds
* You are pregnant or lactating
* You have high blood pressure (greater than 159 mmHg systolic or 99 mmHg diastolic).
* You use tobacco or other nicotine products
* You have a medical condition or take medications that influence heart rate or metabolic rate (for example - beta blockers, antihistamines, anti-depressants, diuretics, thyroid medications).
* You have physical limitations that prevent performance of pedal motions or normal walking. You have any previous history of, or clinical symptoms or signs of, cardiovascular disease, stroke or transient ischemic attacks (TIAs), chest pain, unusual shortness of breath during physical activity, severe ankle edema (swelling), or intermittent claudication (pain caused by lack of blood flow during physical activity).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure | Cross-sectional; single visit
  Energy expenditure will be measured using a portable metabolic system while performing common office tasks or desk work while sitting, standing, and walking. The portable metabolic system consists of a small gas analysis unit and a battery positioned on the abdomen and mid-back, respectively. Respiratory gases are collected by mask that fits over the mouth and nose and analyzed by the unit. The mask does not restrict a participant's breathing, vision or line of sight.

SECONDARY OUTCOMES:
Heart rate | Cross-sectional; single visit
  A heart rate monitor will be fastened around their chest using an elastic strap.
Workload (watts) during seated cycling condition | Cross-sectional; single visit
  Participants will be instructed to maintain their preferred pedaling rate during cycling for 10 minutes. Pedal force will be recoreded by specialized pedals.
Speed during treadmill walking condition | Cross-sectional; single visit
  Participants will be instructed to maintain their preferred treadmill speed during treadmill walking for 10 minutes. Speed will be recoreded by someone outside the immediate study group.
Typing accuracy | Cross-sectional, single visit

CONTACTS AND LOCATIONS:
Overall Officials: Neil M Johannsen, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States